CLINICAL TRIAL: NCT00253123
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Risperidone for Treatment of Behavioral Disturbances in Subjects With Dementia
Brief Title: A Study of the Effectiveness and Safety of Risperidone Versus Placebo in the Treatment of Behavioral Disturbances in Patients With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006022
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular
Keywords: Dementia; Alzheimer's disease; vascular dementia; mixed dementia; risperidone; nursing home
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Mixed Dementias | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of risperidone (an antipsychotic medication) versus placebo in the treatment of behavioral disturbances associated with dementia.

DETAILED DESCRIPTION:
Dementia is a term used for a collection of symptoms that can be caused by a number of diseases or injuries that affect the brain. Individuals with dementia have a loss of cognitive function (thinking, perception, learning, verbal communication, memory, judgment), which may lead to behavioral and personality changes (for example, agitation, delusions, hallucinations). Some causes of dementia are reversible; however, irreversible dementia is caused by certain conditions, such as Alzheimer's disease. Dementia is common in elderly individuals, but it is not a normal part of aging. This is a randomized, double-blind, parallel-group, placebo-controlled study comparing the effectiveness and safety of risperidone to placebo in patients with behavioral disturbances associated with dementia. The study is composed of a screening visit, followed by two study phases: a 1-week run-in period in which patients are discontinued from other antipsychotic drugs and receive placebo twice daily, and a 12-week double-blind period. At the end of the run-in period, patients are randomly assigned to one of three risperidone doses (0.5, 1, or 2 mg/day) or placebo. All patients randomized to risperidone start with 0.25 mg twice daily. During the first week of the double-blind period, patients assigned to the 1 mg/day dose group have their doses increased to 0.5 mg twice daily and patients assigned to the 2 mg/day dose group have their doses increased to 1 mg twice daily. These three assigned doses continue for an additional 11 weeks. The primary measure of effectiveness is the change from baseline in the clinical response, defined as a reduction of >= 30% from baseline on the total Behavior Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD) score. Additional efficacy testing includes the Clinical Global Impressions (CGI), a rating system used to evaluate the overall and severity of clinical change in a patient with various diseases affecting the brain; the Cohen-Mansfield Agitation Inventory (CMAI), a questionnaire evaluating agitation that is completed by the patient's caregiver; the Physical Self-Maintenance Scale (PSMS), a scale that measures activities of daily living (for example, toileting, dressing, grooming, feeding, etc.). Safety evaluations include the incidence of adverse events; results of clinical laboratory tests (hematology, biochemistry, urinalysis); measurements of vital signs; physical examination and electrocardiogram (ECG) findings; and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that risperidone is more effective than placebo, as measured by a change from baseline on the total BEHAVE-AD score, in treating behavioral disturbances in demented patients. Risperidone tablets (or placebo tablets) taken orally, starting with 0.25 mg twice daily, continuing at this dose for the 0.25 twice daily group and gradually increasing to either 0.5 mg twice daily or 1 mg twice daily in the other risperidone dose groups. Treatment duration is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of dementia of the Alzheimer's type, mixed dementia, or vascular dementia, as classified by the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* a score of 4 or more on the Functional Assessment Staging (FAST), a diagnostic tool for determining the stage of dementia
* a score of 23 or lower on the Mini-Mental State Examination (MMSE), a clinical measure used to evaluate cognition
* a BEHAVE-AD total score of at least 8, and a BEHAVE-AD global rating of at least 1
* residence in a psychiatric hospital, nursing home, or other long-term care facility for at least 1 month.

Exclusion Criteria:

* Patients with untreated, reversible causes of dementia
* with general medical or neurological conditions in which cognition is diminished (for example, untreated vitamin deficiency, severe liver or kidney malfunctions, brain tumor, etc.)
* with dementia related to HIV infection (human immunodeficiency virus)
* with a substance-induced persisting dementia
* with psychiatric disorders that could account for the behavior disturbances, such as schizophrenia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Study Completion 1997-03 (Actual)

PRIMARY OUTCOMES:
Reduction of >= 30% from baseline to the end of double-blind treatment on the total BEHAVE-AD score.

SECONDARY OUTCOMES:
Change from baseline to the end of double-blind treatment in BEHAVE-AD global rating and total score; total CMAI score; CGI and CGI change from baseline; PSMS; safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- [Result] Katz IR, Jeste DV, Mintzer JE, Clyde C, Napolitano J, Brecher M. Comparison of risperidone and placebo for psychosis and behavioral disturbances associated with dementia: a randomized, double-blind trial. Risperidone Study Group. J Clin Psychiatry. 1999 Feb;60(2):107-15. doi: 10.4088/jcp.v60n0207. PMID 10084637